CLINICAL TRIAL: NCT06870253
Title: Prospective Evaluation of Bladder CARE™ Assay Utility for the Diagnosis of Bladder Cancer in Patients With Atypical Cytology or Equivocal Cystoscopy
Brief Title: Evaluating Bladder CARE™, a New Non-Invasive Urine Test, for Bladder Cancer Detection in Inconclusive Cases
Status: Active, not recruiting | Type: Observational
Sponsor: Pangea Laboratory LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: PAN001-24 BCA
Record Dates: First submitted 2025-03-05; First posted 2025-03-11 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Bladder Cancer; Urothelial Carcinoma Bladder
Keywords: Bladder CARE™; Bladder Cancer; Atypical Cytology; Equivocal Cystoscopy; Bladder Cancer Detection; Hematuria; Non-Invasive Urine Test; Urological; Urology; Microhematuria; Gross Hematuria; Urothelial Carcinoma; Bladder Cancer Biomarkers; Urinary Biomarker; Urologic Oncology; Inconclusive Cystoscopy Results; Inconclusive Cytology Results; Urine-Based Bladder Cancer Detection
MeSH Terms: conditions — Urinary Bladder Neoplasms; Hematuria; Carcinoma, Transitional Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

SUMMARY:
The goal of this observational study is to learn about the performance of the Bladder CARE™ Assay in patients suspected of having bladder cancer with atypical cytology or equivocal cystoscopy results. The main question it aims to answer is:

• Does the Bladder CARE™ Assay detect bladder cancer in patients who have inconclusive cytology or cystoscopy results?

Participants will provide one voided urine specimen on the day of, and prior to, the routine, scheduled standard of care initial or repeat cystoscopy procedure. A medical records review will occur at two follow-up timepoints, (6 months and 12 months after the urine specimen collection), to document oncology-urinary-related clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years of age at time of informed consent.
2. Subject or the subject's legally authorized representative provides written informed consent.
3. Subject is willing to follow all study procedures and available for the duration of the study.
4. Patients with atypical cytology or equivocal cystoscopy results within 3 months before screening.
5. Subject is scheduled for initial or repeat cystoscopy, with or without pathology.
6. Subject is willing to provide one voided urine specimen of at least 80 ml on the same day, but prior to scheduled initial or repeat cystoscopy, with or without pathology.

Exclusion Criteria:

1. Pregnant or planning to become pregnant at the time of screening.
2. Positive cystoscopy within 3 months of screening indicating presence of bladder cancer.
3. Genitourinary manipulation (flexible or rigid cystoscopy, catheterization, urethral dilation, URS, ureteral stent) within 14 days before urine specimen collection.
4. History of augmentation cystoplasty.
5. History of continent cutaneous diversion or ileal conduit.
6. History of orthotopic bladder substitution or orthotopic neobladder.
7. Concomitant use of an investigational drug which has been administered or may be administered within the 30 days leading up to providing informed consent or may be administered through the time of urine specimen.
8. New or recurrent NMIBC (non-muscle invasive bladder cancer) diagnosis within three months of study enrollment.
9. An active malignancy (bladder or other) diagnosis within 3 months of study enrollment.
10. Patients with a history of NMIBC have undergone intravesical or infusion therapy and completed treatment less than 6 weeks prior to study enrollment.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Urology practice
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-06-03 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Evaluate Bladder CARE™ Assay performance for detecting bladder cancer in patients with atypical cytology or equivocal cystoscopy | From enrollment to the end of the study at 12 months
  Assess the sensitivity, specificity, positive predictive value (PPV), and negative predictive value (NPV), of the Bladder CARE™ Assay to the gold standard diagnostic methods for detecting bladder cancer in patients with atypical cytology or equivocal cystoscopy results.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey R. Karnes, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
This IPD sharing plan entails sharing de-identified individual participant data (IPD) exclusively through the publication of results from this clinical trial in a reputable medical journal. The shared data will include essential de-identified demographic information such as age, gender, race/ethnicity, clinical outcomes and summary results. Additionally, the performance metrics of the Bladder CARE™ Assay will be disclosed, providing insights into its effectiveness and utility in clinical settings.
  By disseminating this information through a peer-reviewed journal, we aim to contribute to the scientific community's understanding of the Bladder CARE™ Assay and its implications for patient care, while ensuring that the data is contextualized within the scope of our research findings. This approach aligns with our commitment to transparency and the advancement of medical knowledge. Once accepted, the article will be published.
Time Frame: Beginning 1 year after publication with no end date
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee and a signed data use agreement